CLINICAL TRIAL: NCT00342641
Title: Associations of Hematologic Malignancies and Thyroid Cancer With HCV Infection Among US Military Veterans
Brief Title: Association Between Hepatitis C Virus Infection and Hematologic and Thyroid Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905172; 05-C-N172
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-13

CONDITIONS: Hepatitis C Virus
Keywords: Lymphoma; Multiple Myeloma; Thyroiditis; Cohort Study; Record linkage study; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Lymphoma; Multiple Myeloma; Thyroiditis

SUMMARY:
This study will investigate the possible relationship between infection with hepatitis C virus (HCV) and the development of certain hematologic cancers (Non-Hodgkin's lymphoma, Hodgkin's lymphoma, chronic lymphocytic leukemia, multiple myeloma) and thyroid cancer. HCV causes chronic hepatitis, cirrhosis, and liver cancer. It is transmitted primarily through injection drug use and transfusion of infected blood. Studies have shown that HCV may also be linked to hematologic cancers and thyroid cancer.

This retrospective study will examine medical records from veterans with and without HCV infection who previously received treatment in the Veterans Administration medical system. Data collected on each subject will include the subject's race, sex, age and era of military service, presence of liver disease or thyroiditis at their baseline clinic visit, number of inpatient visits in the past 5 years and outpatient visits in the past year, and the presence of various specified cancers. The prevalence of cancer and other conditions among HCV-infected subjects and non-HCV infected subjects at baseline and the subsequent development of the cancers of interest in these two groups will be compared and analyzed for a possible causal relationship.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) may be a cause of hematologic malignancies and thyroid cancer. HCV infection is common among U.S. military veterans receiving care in the Veterans Administration healthcare system. The investigators propose a retrospective cohort study using VA administrative databases. A cohort of approximately 147,000 HCV-infected veterans has been identified for the period 1997-2004. Likewise, a cohort of approximately 573,000 HCV-uninfected veterans has been identified for the same period. These subjects are being evaluated for the diagnosis of hematologic malignancies, thyroid cancer, and related medical conditions as recorded in VA databases. The comparison of the prevalence and incidence of these cancers in the two cohorts will provide a test of the hypothesis that HCV infection can cause these cancers.

The investigators will also evaluate the association between HCV infection and several other medical conditions, which might be related to HCV infection, specifically: immune thrombocytopenic purpura, autoimmune hemolytic anemia, cholangiocarcinoma, cholangitis, and pancreatic cancer.

ELIGIBILITY:
* None given.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 815000 (Estimated)
Dates: Start 2005-06-08; Study Completion 2011-12-13

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Veterans AFfairs Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Dominitz JA, Boyko EJ, Koepsell TD, Heagerty PJ, Maynard C, Sporleder JL, Stenhouse A, Kling MA, Hrushesky W, Zeilman C, Sontag S, Shah N, Ona F, Anand B, Subik M, Imperiale TF, Nakhle S, Ho SB, Bini EJ, Lockhart B, Ahmad J, Sasaki A, van der Linden B, Toro D, Martinez-Souss J, Huilgol V, Eisen S, Young KA. Elevated prevalence of hepatitis C infection in users of United States veterans medical centers. Hepatology. 2005 Jan;41(1):88-96. doi: 10.1002/hep.20502. PMID 15619249
- [Background] Engels EA, Chatterjee N, Cerhan JR, Davis S, Cozen W, Severson RK, Whitby D, Colt JS, Hartge P. Hepatitis C virus infection and non-Hodgkin lymphoma: results of the NCI-SEER multi-center case-control study. Int J Cancer. 2004 Aug 10;111(1):76-80. doi: 10.1002/ijc.20021. PMID 15185346
- [Background] Negri E, Little D, Boiocchi M, La Vecchia C, Franceschi S. B-cell non-Hodgkin's lymphoma and hepatitis C virus infection: a systematic review. Int J Cancer. 2004 Aug 10;111(1):1-8. doi: 10.1002/ijc.20205. PMID 15185336